CLINICAL TRIAL: NCT00525512
Title: A Randomized, Double-blind, Placebo-controlled Two-year Trial to Examine the Changes in Exercise Endurance and COPD Treated With Tiotropium Once Daily (EXACTT)
Brief Title: Tiotropium In Exercise
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.368; 2006-004610-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Results first posted 2011-09-23 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Tiotropium Bromide

ARMS (2):
- tiotropium 18mcg (Experimental): Oral inhalation once daily of 18mcg tiotropium via handihaler
  Interventions: Drug: tiotropium 18 mcg
- Placebo (Placebo Comparator): Oral inhalation once daily of placebo matching tiotropium via handihaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tiotropium 18 mcg — Oral inhalation once daily of 18mcg tiotropium via handihaler
  Arms: tiotropium 18mcg
Drug: Placebo — Oral inhalation of once-daily placebo matching tiotropium via handihaler
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effects on exercise duration of 96 weeks treatment with 18 mcg tiotropium (Spiriva HandiHaler) daily as compared to placebo, in patients with COPD.

ELIGIBILITY:
Inclusion criteria

1. All patients must sign an informed consent
2. Diagnosis of COPD with specific spirometric criteria (determined at study visits)
3. Age >= 40 years
4. Medical Research Council Dyspnoea score >= 2
5. Current or ex-smoker with a >= 10 pack-year smoking history
6. Ability to exercise on treadmill

Exclusion criteria

1. Significant diseases other than COPD such as history of life-threatening pulmonary obstruction, thoracotomy with pulmonary resection, interstitial lung disease, CF, pulmonary thromboembolic disease, clinically evident bronchiectasis, active tuberculosis, or known moderate to severe renal impairment
2. Clinical history of asthma
3. Use of supplemental oxygen therapy
4. Respiratory tract infection or COPD exacerbation in the 6 weeks prior to Visit 1 or during the washout period prior to Visit 3 (may randomize 6 weeks after recovery)
5. Recent history (<= 12 months) of myocardial infarction
6. Unstable or life-threatening cardiac arrhythmia
7. Malignancy treated with radiation therapy or chemotherapy in the last 5 years
8. Pregnant or nursing women
9. Known hypersensitivity to anticholinergic drugs or any component of the study medications
10. Participation in pulmonary or cardiac rehab program within 13 weeks of Visit 1
11. Estimated life expectancy < 2 years
12. Symptomatic prostatic hyperplasia or bladder neck obstruction
13. Known narrow-angle glaucoma
14. Any condition that is contraindicated for exercise
15. Orthopaedic, muscular, neurological or cardiac disease that would interfere with regular participation in aerobic exercise or with exercise testing
16. Body mass index < 18 kg/m2 or >35 kg/m2 list truncated for space

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (62):
- United States (21):
  - 205.368.01023 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 205.368.01022 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 205.368.01003 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.368.01008 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 205.368.01017 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 205.368.01028 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 205.368.01004 Boehringer Ingelheim Investigational Site, Bay Pines, Florida
  - 205.368.01013 Boehringer Ingelheim Investigational Site, North Miami Beach, Florida
  - 205.368.01025 Boehringer Ingelheim Investigational Site, Hazard, Kentucky
  - 205.368.01029 Boehringer Ingelheim Investigational Site, Biddeford, Maine
  - 205.368.01016 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 205.368.01002 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 205.368.01021 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 205.368.01014 Boehringer Ingelheim Investigational Site, Albany, New York
  - 205.368.01030 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 205.368.01018 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.368.01027 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 205.368.01019 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 205.368.01020 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 205.368.01024 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 205.368.01015 Boehringer Ingelheim Investigational Site, Dallas, Texas
- Argentina (2):
  - 205.368.54001 Boehringer Ingelheim Investigational Site, Rosario
  - 205.368.54002 Boehringer Ingelheim Investigational Site, Vicente López
- Brazil (3):
  - 205.368.55003 Boehringer Ingelheim Investigational Site, Goiânia
  - 205.368.55004 Boehringer Ingelheim Investigational Site, Porto Alegre - RS
  - 205.368.55002 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (6):
  - 205.368.07006 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 205.368.07001 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 205.368.07003 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 205.368.07004 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 205.368.07005 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 205.368.07008 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Germany (6):
  - 205.368.49005 Boehringer Ingelheim Investigational Site, Berlin
  - 205.368.49003 Boehringer Ingelheim Investigational Site, Cologne
  - 205.368.49004 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 205.368.49006 Boehringer Ingelheim Investigational Site, Münster
  - 205.368.49002 Boehringer Ingelheim Investigational Site, Schmallenberg
  - 205.368.49001 Boehringer Ingelheim Investigational Site, Tübingen
- Italy (4):
  - 205.368.39006 Boehringer Ingelheim Investigational Site, Ferrara
  - 205.368.39004 Boehringer Ingelheim Investigational Site, Milan
  - 205.368.39002 Boehringer Ingelheim Investigational Site, Parma
  - 205.368.39001 Boehringer Ingelheim Investigational Site, Pisa
- Portugal (2):
  - 205.368.35103 Boehringer Ingelheim Investigational Site, Coimbra
  - 205.368.35102 Boehringer Ingelheim Investigational Site, Matosinhos Municipality
- Russia (5):
  - 205.368.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 205.368.70004 Boehringer Ingelheim Investigational Site, Moscow
  - 205.368.70005 Boehringer Ingelheim Investigational Site, Moscow
  - 205.368.70006 Boehringer Ingelheim Investigational Site, Moscow
  - 205.368.70007 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Spain (6):
  - 205.368.34005 Hospital Germans Trias i Pujol, Badalona (Barcelona)
  - 205.368.34002 Hospital de Cruces, Barakaldo (Bilbao)
  - 205.368.34001 Hospital Clinic i Provincial de Barcelona, Barcelona
  - 205.368.34003 Hospital Gregorio Maranon, Madrid
  - 205.368.34004 Hospital Universitario Vírgen del Rocío, Seville
  - 205.368.34006 Boehringer Ingelheim Investigational Site, Seville
- Taiwan (4):
  - 205.368.88604 Boehringer Ingelheim Investigational Site, Keelung
  - 205.368.88602 Boehringer Ingelheim Investigational Site, Taichung
  - 205.368.88603 Boehringer Ingelheim Investigational Site, Taipei
  - 205.368.88601 Chang Gung Memorial Hosp-Linkou, Taoyuan District
- Ukraine (3):
  - 205.368.38003 Boehringer Ingelheim Investigational Site, Dnyepropyetrovsk
  - 205.368.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 205.368.38002 Boehringer Ingelheim Investigational Site, Kiev

REFERENCES:
- [Derived] Cooper CB, Celli BR, Jardim JR, Wise RA, Legg D, Guo J, Kesten S. Treadmill endurance during 2-year treatment with tiotropium in patients with COPD: a randomized trial. Chest. 2013 Aug;144(2):490-497. doi: 10.1378/chest.12-2613. PMID 23558890

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- Tiotropium: Patients randomized to treatment with Tiotropium 18 micrograms
- Placebo / Open Tiotropium: Patients receive open label tiotropium following placebo
- Tiotropium / Open Tiotropium: Patients receive open label tiotropium following tiotropium
Period: Double-Blind Phase
Arm/Group | Placebo | Tiotropium | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Started | 259 | 260 | 0 | 0
Completed | 163 | 194 | 0 | 0
Not Completed | 96 | 66 | 0 | 0
Not completed — Adverse Event | 48 | 28 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 12 | 0 | 0
Not completed — Lack of Efficacy | 13 | 5 | 0 | 0
Not completed — Other reason (not specified) | 12 | 13 | 0 | 0
Period: Open-Label Phase
Arm/Group | Placebo | Tiotropium | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Started | 0 | 0 | 164 | 194
Completed | 0 | 0 | 158 | 189
Not Completed | 0 | 0 | 6 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Other reason (not specified) | 0 | 0 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tiotropium | Total
Number analyzed (Participants) | 259 | 260 | 519
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.5) | 64.7 (8.2) | 64.6 (8.3)
Age, Customized [Number; unit: participants]
  <= 55 | 37 | 38 | 75
  > 55 to <= 65 | 101 | 93 | 194
  > 65 | 121 | 129 | 250
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 61 | 118
  Male | 202 | 199 | 401
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian / Alaskan Native | 2 | 2 | 4
  Asian | 14 | 22 | 36
  Black / African American | 6 | 10 | 16
  Hawaiian / Pacific Islander | 0 | 0 | 0
  White | 237 | 226 | 463
Smoking Status [Number; unit: participants]
  Never smoked | 0 | 0 | 0
  Ex-smoker | 174 | 169 | 343
  Currently smokes | 85 | 91 | 176
Smoking history [Mean (Standard Deviation); unit: pack years] | 51.04 (26.29) | 52.15 (28.95) | 51.6 (27.64)
Duration of COPD (Chronic Obstructive Pulmonary Disease) [Mean (Standard Deviation); unit: years] | 8.80 (6.99) | 8.70 (6.27) | 8.75 (6.63)
Height [Mean (Standard Deviation); unit: centimeters] | 169.6 (8.5) | 169.7 (9.2) | 169.7 (8.9)
Weight [Mean (Standard Deviation); unit: kilograms] | 77.4 (15.0) | 75.4 (16.0) | 76.4 (15.5)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kilograms / square meter] | 26.8 (4.23) | 26.0 (4.38) | 26.4 (4.31)
Alcohol status [Number; unit: participants]
  Non drinker | 114 | 123 | 237
  Drinks - no interference with study | 145 | 137 | 282
  Drinks - possible interference with study | 0 | 0 | 0
LABA (Long Acting Beta Agonist) use at randomization [Number; unit: participants]
  No | 104 | 107 | 211
  Yes | 155 | 153 | 308
ICS (Inhaled Cortico Steroid) use at randomization [Number; unit: participants]
  No | 108 | 101 | 209
  Yes | 151 | 159 | 310
LABA / ICS use at randomization [Number; unit: participants]
  No | 133 | 131 | 264
  Yes | 126 | 129 | 255
Anticholinergic use at screening [Number; unit: participants]
  No | 139 | 139 | 278
  Yes | 120 | 121 | 241

OUTCOME MEASURES:

1. Primary Outcome: 90% Constant Work Rate (CWR) Treadmill Endurance Time at 96 Weeks - Double-Blind Phase
Description: Efficacy was assessed by measuring the exercise duration during a treadmill exercise test.
Time Frame: baseline, 96 weeks
Population: Full Analysis Set (FAS) includes all treated participants with a baseline and any post-dosing exercise duration data
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
seconds | 297.1 [265.0 to 333.0] | 336.6 [302.5 to 374.7]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.1062, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Adjusted mean ratio = 1.13, 95% CI [0.97 to 1.32]

2. Secondary Outcome: 90% Constant Work Rate (CWR) Treadmill Endurance Time at 8 Weeks - Double-Blind Phase
Description: Efficacy was assessed by measuring the exercise duration during a treadmill exercise test.
Time Frame: baseline, 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
seconds | 304.9 [284.7 to 326.5] | 343.0 [321.2 to 366.2]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Adjusted mean ratio = 1.12, 95% CI [1.03 to 1.23]

3. Secondary Outcome: 90% Constant Work Rate (CWR) Treadmill Endurance Time at 16 Weeks - Double-Blind Phase
Description: Efficacy was assessed by measuring the exercise duration during a treadmill exercise test.
Time Frame: baseline, 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
seconds | 308.6 [286.2 to 332.8] | 338.6 [315.2 to 363.7]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0597, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Adjusted mean ratio = 1.10, 95% CI [1.00 to 1.21]

4. Secondary Outcome: 90% Constant Work Rate (CWR) Treadmill Endurance Time at 32 Weeks - Double-Blind Phase
Description: Efficacy was assessed by measuring the exercise duration during a treadmill exercise test.
Time Frame: baseline, 32 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
seconds | 311.8 [286.3 to 339.5] | 358.7 [330.9 to 388.9]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0131, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Adjusted mean ratio = 1.15, 95% CI [1.03 to 1.29]

5. Secondary Outcome: 90% Constant Work Rate (CWR) Treadmill Endurance Time at 48 Weeks - Double-Blind Phase
Description: Efficacy was assessed by measuring the exercise duration during a treadmill exercise test.
Time Frame: baseline, 48 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
seconds | 309.8 [284.0 to 337.9] | 365.7 [336.8 to 397.0]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Adjusted mean ratio = 1.18, 95% CI [1.05 to 1.32]

6. Secondary Outcome: 90% Constant Work Rate (CWR) Treadmill Endurance Time at 64 Weeks - Double-Blind Phase
Description: Efficacy was assessed by measuring the exercise duration during a treadmill exercise test.
Time Frame: baseline, 64 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
seconds | 313.4 [284.7 to 344.9] | 349.0 [318.7 to 382.2]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0945, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Adjusted mean ratio = 1.11, 95% CI [0.98 to 1.26]

7. Secondary Outcome: 90% Constant Work Rate (CWR) Treadmill Endurance Time at 80 Weeks - Double-Blind Phase
Description: Efficacy was assessed by measuring the exercise duration during a treadmill exercise test.
Time Frame: baseline, 80 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
seconds | 302.8 [273.5 to 335.2] | 340.1 [309.0 to 374.4]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0899, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Adjusted mean ratio = 1.12, 95% CI [0.98 to 1.28]

8. Secondary Outcome: Pre-treatment Forced Expiratory Volume in 1 Second (FEV1) at 8 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 8 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.082 (0.017) | 1.198 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.116, 95% CI [0.073 to 0.160]

9. Secondary Outcome: Pre-treatment Forced Expiratory Volume in 1 Second (FEV1) at 16 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 16 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.082 (0.018) | 1.164 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.082, 95% CI [0.036 to 0.128]

10. Secondary Outcome: Pre-treatment Forced Expiratory Volume in 1 Second (FEV1) at 32 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 32 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.090 (0.019) | 1.179 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.089, 95% CI [0.041 to 0.137]

11. Secondary Outcome: Pre-treatment Forced Expiratory Volume in 1 Second (FEV1) at 48 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 48 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.066 (0.019) | 1.172 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.105, 95% CI [0.058 to 0.153]

12. Secondary Outcome: Pre-treatment Forced Expiratory Volume in 1 Second (FEV1) at 64 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 64 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.066 (0.020) | 1.157 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.090, 95% CI [0.040 to 0.141]

13. Secondary Outcome: Pre-treatment Forced Expiratory Volume in 1 Second (FEV1) at 80 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 80 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.039 (0.019) | 1.134 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Median Difference (Final Values) = 0.094, 95% CI [0.045 to 0.144]

14. Secondary Outcome: Pre-treatment Forced Expiratory Volume in 1 Second (FEV1) at 96 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.050 (0.021) | 1.125 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0059, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.075, 95% CI [0.022 to 0.128]

15. Secondary Outcome: Post-treatment Forced Expiratory Volume in 1 Second (FEV1) at 8 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 8 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.126 (0.017) | 1.280 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.154, 95% CI [0.110 to 0.198]

16. Secondary Outcome: Post-treatment Forced Expiratory Volume in 1 Second (FEV1) at 16 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 16 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.092 (0.017) | 1.254 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.162, 95% CI [0.117 to 0.208]

17. Secondary Outcome: Post-treatment Forced Expiratory Volume in 1 Second (FEV1) at 32 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 32 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.113 (0.018) | 1.259 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.145, 95% CI [0.099 to 0.192]

18. Secondary Outcome: Post-treatment Forced Expiratory Volume in 1 Second (FEV1) at 48 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 48 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.105 (0.019) | 1.232 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.127, 95% CI [0.077 to 0.176]

19. Secondary Outcome: Post-treatment Forced Expiratory Volume in 1 Second (FEV1) at 64 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 64 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.097 (0.020) | 1.230 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.134, 95% CI [0.083 to 0.185]

20. Secondary Outcome: Post-treatment Forced Expiratory Volume in 1 Second (FEV1) at 80 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 80 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.079 (0.020) | 1.228 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.149, 95% CI [0.097 to 0.202]

21. Secondary Outcome: Post-treatment Forced Expiratory Volume in 1 Second (FEV1) at 96 Weeks - Double-Blind Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 1.072 (0.021) | 1.202 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.130, 95% CI [0.077 to 0.183]

22. Secondary Outcome: Pre-treatment Forced Vital Capacity (FVC) at 8 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 8 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.432 (0.035) | 2.649 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.217, 95% CI [0.127 to 0.307]

23. Secondary Outcome: Pre-treatment Forced Vital Capacity (FVC) at 16 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 16 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.407 (0.038) | 2.564 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.157, 95% CI [0.058 to 0.255]

24. Secondary Outcome: Pre-treatment Forced Vital Capacity (FVC) at 32 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 32 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.425 (0.040) | 2.607 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.182, 95% CI [0.078 to 0.286]

25. Secondary Outcome: Pre-treatment Forced Vital Capacity (FVC) at 48 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 48 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.406 (0.041) | 2.640 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.234, 95% CI [0.130 to 0.339]

26. Secondary Outcome: Pre-treatment Forced Vital Capacity (FVC) at 64 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 64 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.423 (0.046) | 2.584 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.161, 95% CI [0.040 to 0.281]

27. Secondary Outcome: Pre-treatment Forced Vital Capacity (FVC) at 80 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 80 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.343 (0.042) | 2.555 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.212, 95% CI [0.102 to 0.322]

28. Secondary Outcome: Pre-treatment Forced Vital Capacity (FVC) at 96 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.368 (0.044) | 2.609 (0.041)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.241, 95% CI [0.128 to 0.355]

29. Secondary Outcome: Post-treatment Forced Vital Capacity (FVC) at 8 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 8 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.529 (0.038) | 2.806 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.277, 95% CI [0.179 to 0.375]

30. Secondary Outcome: Post-treatment Forced Vital Capacity (FVC) at 16 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 16 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.442 (0.039) | 2.767 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.325, 95% CI [0.226 to 0.425]

31. Secondary Outcome: Post-treatment Forced Vital Capacity (FVC) at 32 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 32 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.462 (0.042) | 2.816 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.353, 95% CI [0.245 to 0.461]

32. Secondary Outcome: Post-treatment Forced Vital Capacity (FVC) at 48 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 48 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.499 (0.041) | 2.758 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.259, 95% CI [0.154 to 0.365]

33. Secondary Outcome: Post-treatment Forced Vital Capacity (FVC) at 64 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 64 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.466 (0.041) | 2.767 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.300, 95% CI [0.194 to 0.406]

34. Secondary Outcome: Post-treatment Forced Vital Capacity (FVC) at 80 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 80 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.479 (0.043) | 2.733 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.254, 95% CI [0.144 to 0.364]

35. Secondary Outcome: Post-treatment Forced Vital Capacity (FVC) at 96 Weeks - Double-Blind Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 224 | 238
liters | 2.420 (0.048) | 2.753 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.333, 95% CI [0.209 to 0.456]

36. Secondary Outcome: Borg Scale of Dyspnea at Isotime After 96 Weeks - Double-Blind Phase
Description: Borg scale assessed degreee of discomfort on a scale from 0 (Nothing at all) to 10 (Maximal)
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 162 | 193
units on scale | 4.1 (0.16) | 3.8 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.1131, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = -0.32, 95% CI [-0.72 to 0.08]

37. Secondary Outcome: Borg Scale of Peak Dyspnea After 96 Weeks - Double-Blind Phase
Description: Borg scale assessed degreee of discomfort on a scale from 0 (Nothing at all) to 10 (Maximal)
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: unit on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
unit on scale | 5.6 (0.14) | 5.6 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.9071, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = -0.02, 95% CI [-0.38 to 0.33]

38. Secondary Outcome: Borg Scale of Peak Leg Discomfort After 96 Weeks - Double-Blind Phase
Description: Borg scale assessed degreee of discomfort on a scale from 0 (Nothing at all) to 10 (Maximal)
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: unit on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
unit on scale | 4.0 (0.18) | 4.1 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.6878, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.09, 95% CI [-0.35 to 0.53]

39. Secondary Outcome: Change From Baseline in Physician Global Evaluation at 8 Weeks - Double-Blind Phase
Description: The evaluation represented the global opinion of the overall clinical condition on a scale of: 1-2 (Poor), 3-4 (Fair), 5-6 (Good), 7-8 (Excellent)
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Error); unit: unit on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
unit on scale | -0.04 (0.999) | 0.32 (0.986)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.36, 95% CI [-2.39 to 3.11]

40. Secondary Outcome: Change From Baseline in Physician Global Evaluation at 16 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 16 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | 0.02 (1.068) | 0.35 (1.083)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.33, 95% CI [-2.66 to 3.31]

41. Secondary Outcome: Change From Baseline in Physician Global Evaluation at 32 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 32 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | -0.04 (1.153) | 0.30 (1.186)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.34, 95% CI [-2.91 to 3.58]

42. Secondary Outcome: Change From Baseline in Physician Global Evaluation at 48 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 48 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | 0.03 (1.143) | 0.25 (1.165)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.23, 95% CI [-2.97 to 3.43]

43. Secondary Outcome: Change From Baseline in Physician Global Evaluation at 64 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 64 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | 0.03 (1.168) | 0.25 (1.170)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.22, 95% CI [-3.02 to 3.46]

44. Secondary Outcome: Change From Baseline in Physician Global Evaluation at 80 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 80 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | -0.06 (1.217) | 0.10 (1.132)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.16, 95% CI [-3.10 to 3.41]

45. Secondary Outcome: Change From Baseline in Physician Global Evaluation at 96 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 96 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | -0.07 (1.222) | 0.10 (1.220)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.17, 95% CI [-3.22 to 3.55]

46. Secondary Outcome: Change From Baseline in Patient Global Evaluation at 8 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | -0.03 (1.134) | 0.34 (1.138)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.37, 95% CI [-2.78 to 3.52]

47. Secondary Outcome: Change From Baseline in Patient Global Evaluation at 16 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 16 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | 0.07 (1.206) | 0.30 (1.159)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.23, 95% CI [-3.05 to 3.51]

48. Secondary Outcome: Change From Baseline in Patient Global Evaluation at 32 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 32 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | 0.13 (1.281) | 0.20 (1.225)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.08, 95% CI [-3.40 to 3.55]

49. Secondary Outcome: Change From Baseline in Patient Global Evaluation at 48 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 48 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | 0.02 (1.365) | 0.18 (1.349)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.15, 95% CI [-3.61 to 3.92]

50. Secondary Outcome: Change From Baseline in Patient Global Evaluation at 64 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 64 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | -0.02 (1.250) | 0.16 (1.424)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.18, 95% CI [-3.53 to 3.90]

51. Secondary Outcome: Change From Baseline in Patient Global Evaluation at 80 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 80 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | -0.08 (1.284) | 0.09 (1.269)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.18, 95% CI [-3.36 to 3.71]

52. Secondary Outcome: Change From Baseline in Patient Global Evaluation at 96 Weeks - Double-Blind Phase
Description: as for outcome 39
Time Frame: baseline, 96 weeks
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 225 | 239
units on scale | -0.04 (1.455) | 0.03 (1.348)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.07, 95% CI [-3.82 to 3.96]

53. Secondary Outcome: Saint George's Respiratory Questionnaire Total Score at 96 Weeks - Double-Blind Phase
Description: Score summarises the impact of disease on overall health status with zero indicating best health status and 100 indicating worst possible health status.
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 216 | 220
units on scale | 44.5 (1.13) | 40.5 (1.07)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0072, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = -4.03, 95% CI [-6.97 to -1.10]

54. Secondary Outcome: Saint George's Respiratory Questionnaire Activity Component Score at 96 Weeks - Double-Blind Phase
Description: as for outcome 53
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 216 | 220
units on scale | 56.9 (1.39) | 54.6 (1.32)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.2029, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = -2.33, 95% CI [-5.91 to 1.26]

55. Secondary Outcome: Saint George's Respiratory Questionnaire Impact Component Score at 96 Weeks - Double-Blind Phase
Description: as for outcome 53
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 216 | 220
units on scale | 34.0 (1.25) | 30.4 (1.20)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0313, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = -3.58, 95% CI [-6.84 to -0.32]

56. Secondary Outcome: Saint George's Respiratory Questionnaire Symptoms Component Score at 96 Weeks - Double-Blind Phase
Description: as for outcome 53
Time Frame: baseline, 96 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 216 | 220
units on scale | 54.4 (1.73) | 45.5 (1.63)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — Based on a MMRM analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = -8.94, 95% CI [-13.37 to -4.52]

57. Secondary Outcome: Patients With COPD Exacerbation (Survival Analysis) - Double-Blind Phase
Description: COPD exacerbation is a complex of symptoms related to COPD with a duration of three days or more requiring a change of treatment.
Time Frame: baseline, 96 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 259 | 260
participants
  Patients with exacerbations | 102 | 112
  Censored patients | 157 | 148
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p = 0.6541, Regression, Cox — Based on a MMRM analysis with terms for treatment, centre and baseline; Cox Proportional Hazard = 0.940, 95% CI [0.719 to 1.230]

58. Secondary Outcome: 90% Constant Work Rate (CWR) Treadmill Endurance Time at 100 Weeks - Open-Label Phase
Description: Efficacy was assessed by measuring the exercise duration during a treadmill exercise test.
Time Frame: baseline, 100 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Number analyzed (Participants) | 150 | 178
seconds | 337.25 [297.63 to 382.14] | 358.80 [318.05 to 404.78]
Statistical Analysis 1: Comparison: Placebo / Open Tiotropium vs Tiotropium / Open Tiotropium; Test type: Superiority or Other; p = 0.4443, ANCOVA — Based on a ANCOVA analysis with terms for treatment, centre and baseline; Adjusted mean ratio = 1.06, 95% CI [0.91 to 1.25]

59. Secondary Outcome: Post-treatment Forced Expiratory Volume in 1 Second (FEV1) at 100 Weeks - Open-Label Phase
Description: FEV1 is the maximal amount of air you can forcefully exhale in one second.
Time Frame: baseline, 100 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Number analyzed (Participants) | 154 | 184
liters | 1.23 (0.02) | 1.23 (0.02)
Statistical Analysis 1: Comparison: Placebo / Open Tiotropium vs Tiotropium / Open Tiotropium; Test type: Superiority or Other; p = 0.8644, ANCOVA — Based on a ANCOVA analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.01, 95% CI [-0.05 to 0.06]

60. Secondary Outcome: Post-treatment Forced Vital Capacity (FVC) at 100 Weeks - Open-Label Phase
Description: FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: baseline, 100 weeks
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Number analyzed (Participants) | 154 | 184
liters | 2.72 (0.05) | 2.77 (0.05)
Statistical Analysis 1: Comparison: Placebo / Open Tiotropium vs Tiotropium / Open Tiotropium; Test type: Superiority or Other; p = 0.4277, ANCOVA — Based on a ANCOVA analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.05, 95% CI [-0.07 to 0.17]

61. Secondary Outcome: Saint George's Respiratory Questionnaire Total Score at 100 Weeks - Open-Label Phase
Description: as for outcome 53
Time Frame: baseline, 100 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Number analyzed (Participants) | 145 | 168
units on scale | 39.82 (1.28) | 39.21 (1.21)
Statistical Analysis 1: Comparison: Placebo / Open Tiotropium vs Tiotropium / Open Tiotropium; Test type: Superiority or Other; p = 0.7071, ANCOVA — Based on a ANCOVA analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = -0.61, 95% CI [-3.81 to 2.59]

62. Secondary Outcome: Saint George's Respiratory Questionnaire Activity Component Score at 100 Weeks - Open-Label Phase
Description: as for outcome 53
Time Frame: baseline, 100 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Number analyzed (Participants) | 145 | 168
units on scale | 53.57 (1.57) | 54.46 (1.49)
Statistical Analysis 1: Comparison: Placebo / Open Tiotropium vs Tiotropium / Open Tiotropium; Test type: Superiority or Other; p = 0.6556, ANCOVA — Based on a ANCOVA analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.89, 95% CI [-3.03 to 4.81]

63. Secondary Outcome: Saint George's Respiratory Questionnaire Impact Component Score at 100 Weeks - Open-Label Phase
Description: as for outcome 53
Time Frame: baseline, 100 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Number analyzed (Participants) | 146 | 168
units on scale | 29.65 (1.38) | 29.67 (1.31)
Statistical Analysis 1: Comparison: Placebo / Open Tiotropium vs Tiotropium / Open Tiotropium; Test type: Superiority or Other; p = 0.9896, ANCOVA — Based on a ANCOVA analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = 0.02, 95% CI [-3.44 to 3.48]

64. Secondary Outcome: Saint George's Respiratory Questionnaire Symptoms Component Score at 100 Weeks - Open-Label Phase
Description: as for outcome 53
Time Frame: baseline, 100 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Number analyzed (Participants) | 146 | 169
units on scale | 45.47 (1.94) | 41.14 (1.85)
Statistical Analysis 1: Comparison: Placebo / Open Tiotropium vs Tiotropium / Open Tiotropium; Test type: Superiority or Other; p = 0.0807, ANCOVA — Based on a ANCOVA analysis with terms for treatment, centre and baseline; Mean Difference (Final Values) = -4.33, 95% CI [-9.19 to 0.53]

65. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs and Physical Examination, Including Vital Status
Description: Clinical Relevant Abnormalities for Vital Signs and Physical examination, including vital status. Any new or clinically relevant worsening of baseline conditions was reported as Adverse Events.
Time Frame: From first drug administration until 30 days after last drug administration
Measure: Number; unit: participants
Arm/Group | Placebo | Tiotropium | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Number analyzed (Participants) | 259 | 260 | 164 | 194
participants
  Blood pressure increased | 0 | 2 | 0 | 0
  Heart rate increased | 1 | 1 | 1 | 0
  Oxygen saturation decreased | 1 | 0 | 0 | 0
  Weight decreased | 1 | 2 | 0 | 0
  Fatal | 6 | 6 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration.
Arm/Group | Placebo | Tiotropium | Placebo / Open Tiotropium | Tiotropium / Open Tiotropium
Serious Adverse Events (participants affected / at risk) | 59/259 | 63/260 | 3/164 | 6/194
Other Adverse Events (participants affected / at risk) | 135/259 | 128/260 | 5/164 | 5/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | Tiotropium (N=260) | Placebo / Open Tiotropium (N=164) | Tiotropium / Open Tiotropium (N=194)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Blindness (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 5 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 12 | 11 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 | 21 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 2 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | Tiotropium (N=260) | Placebo / Open Tiotropium (N=164) | Tiotropium / Open Tiotropium (N=194)
Nasopharyngitis (Infections and infestations) | 22 | 12 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 14 | 18 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 14 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 79 | 79 | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 16 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.